CLINICAL TRIAL: NCT06037889
Title: Efficacy and Safety of Tirofiban in Patients With Acute Branch Atheromatous Disease (BAD)- Related Stroke (BRANT)
Brief Title: Efficacy and Safety of Tirofiban for Patients With BAD (BRANT)
Acronym: BRANT
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Pharmaron (Chengdu) Clinical Services Co., Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BAD-RCT202201
Record Dates: First submitted 2023-09-07; First posted 2023-09-14 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-11

CONDITIONS: Branch Atheromatous Disease
Keywords: Branch atheromatous disease; Tirofiban; Stroke; Treatment Outcome; Magnetic Resonance Imaging
MeSH Terms: conditions — Stroke | interventions — Tirofiban; Sodium Chloride; Aspirin; Clopidogrel

STUDY DESIGN:
Intervention Model Description: multi-center, randomized, open label, blinded endpoint, parallel controlled trial
Who Masked: Outcomes Assessor
Masking Description: Our study is an open label, blinded endpoint trail. The primary outcome should be measured in a blinded manner, and the qualified evaluator is defined as: 1) Attending neurologists or above; 2) Complete the training for mRS score before the initiation of patient enrollment; 3) Blind to the antiplatelet treatment of the participants; and 4) Sign the evaluation when it is completed, and inform the other investigators of the results. All the clinical and safety events will be re-examined by the independent Clinical Event Committee (CEC), who are blinded during all procedures.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tirofiban group (Experimental): Intravenous tirofiban will be administered immediately after randomization for a total duration of 48h with a loading dose of 0.4ug/kg/min*30min, followed by a maintenance dose of 0.1ug/kg/min*47.5h.
  Interventions: Drug: Tirofiban
- Standard antiplatelet therapy group (Active Comparator): Standard antiplatelet therapy based on Chinese stroke guideline will be administered after randomization for a total duration of 48h, as the two following types: 1) aspirin 150-300 mg qd, or 2) aspirin 100 mg qd plus clopidogrel 75 mg qd. The time for administration of antiplatelet drugs will be determined by the doctor in conjunction with the participants' use of antiplatelet or anticoagulant medication in the 24h prior to randomization, but the drug should be given as soon as possible after randomization.
  Interventions: Drug: Aspirin tablet; Drug: Clopidogrel tablet

INTERVENTIONS:
Drug: Tirofiban — Tirofiban, a GPIIb/IIIa receptor inhibitor. Intravenous administration.
  Other Names: Tirofiban Hydrochloride and Sodium Chloride Injection
  Arms: Tirofiban group
Drug: Aspirin tablet — Aspirin. Oral administration.
  Arms: Standard antiplatelet therapy group
Drug: Clopidogrel tablet — Clopidogrel. Oral administration.
  Arms: Standard antiplatelet therapy group

SUMMARY:
Branch atheromatous disease (BAD)-related stroke, characterized by subcortical single infarcts without severe stenosis of the large artery, but with a clear atherosclerotic mechanism, is now regarded as a separate stroke type. BAD is associated with early neurological deterioration and poor prognosis, but is lack of effective therapy. The goal of this randomized controlled trial is to test the efficacy and safety of intravenous tirofiban in patients with acute ischemic stroke caused by branch atheromatous disease. The main question it aims to answer is: Compared with standard antiplatelet therapy based on current stroke guideline, whether tirofiban used in acute phase of BAD could improve the proportion of excellent functional outcome (modified Rankin Scale: 0-1) at 90 days. Researcher will also compare the rate of major bleeding between treatment and control groups.

DETAILED DESCRIPTION:
BRANT study is a multicenter, randomized, open label, blinded endpoint, Parallel controlled trial with the primary null hypothesis that, in patients with acute BAD-related stroke, there is no difference in the proportion of excellent outcome in those treated with intravenous Tirofiban compared with those treated with standard antiplatelet therapy based on guideline when subjects are randomized within 48 hours of stroke onset.

The primary objective is to determine whether intravenous tirofiban (a loading dose of 0.4ug/kg/min*30min followed by a maintenance dose of 0.1ug/kg/min*47.5h) is effective in increasing the proportion of excellent functional outcome (mR: 0-1) at 90 days, when initiated within 48 hours of onset. The active comparator is standard antiplatelet therapy based on guideline [ie, 1) aspirin 150-300 mg qd, OR 2) aspirin 100 mg qd plus clopidogrel 75 mg qd] for 48 hours.

Patients with acute BAD-related stroke between 18 and 75 years old, who can be randomized within 48 hours of onset, and meet the BAD Diagnostic Imaging Criteria, will be enrolled. All patients will conduct MRI before randomization.

Subjects will be randomized 1:1 (Tirofiban: Standard antiplatelet therapy). The subjects' eligibility will be assessed by site investigator prior to accessing the Randomization Module, which is generated via the dynamic block randomization method. Only certified and trained personnel can access the randomization website, who will get the information of treatment (ie, Tirofiban or standard antiplatelet therapy) after the subject has be determined eligible.

The treatment period is 48 hours for both study groups. A total of 516 eligible patients will be enrolled. Each participant will be followed for 90 days from randomization. The primary outcome will be assessed by well-trained senior neurologists blinded to the treatment. All the clinical and safety events will be re-examined by the Clinical Event Committee (CEC), who are blinded during all procedures.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-75 years old
2. Acute ischemic stroke
3. Time from onset to randomization ≤48h; if onset time is unknown, time from last known well to randomization ≤48h
4. Meet the following BAD Diagnostic Imaging Criteria

   4.1. DWI infarcts: single (isolated) deep (subcortical) infarcts;

   4.2. The culprit arteries are either Lenticulostriate artery (LSA) or Paramedian pontine artery (PPA), and the infarct lesion on DWI conforms to one of the following characteristics (A/B): A. LSA: 1) "Comma-like" infarct lesions with "Fan-shaped" extension from bottom to top in the coronary position; or 2) ≥ 3 layers (layer thickness 5-7 mm) on axial DWI brain images; B. PPA: The infarct lesion extends from the deep pons to the ventral pons on the axial DWI brain images;

   4.3. No more than 50% stenosis on the parent artery of the criminal artery (i.e. corresponding basilar or middle cerebral artery) (Confirmed by magnetic resonance angiography [MRA] or computed tomography angiography [CTA] or digital substraction angiography [DSA]).
5. Singed informed consent by the patient or legally authorized representatives.

Exclusion Criteria:

1. Transient ischemic attack (TIA)
2. Intracranial hemorrhagic diseases, vascular malformations, aneurysms, brain abscesses, malignant space-occupying lesions, or other non-ischemic intracranial lesions detected by baseline CT/MRI, or MRA/CTA/DSA;
3. Presence of ≥50% stenosis in extracranial artery in tandem relationship ipsilateral to the lesion;
4. Cardiogenic embolism: atrial fibrillation, myocardial infarction, heart valve disease, dilated cardiomyopathy, infective endocarditis, atrioventricular block disease, heart rate less than 50 beats per minute
5. Have received or plan to receive endovascular therapy or thrombolysis after onset;
6. Stroke of other clear causes, e.g., moyamoya disease, arterial entrapment, vasculitis, etc.
7. modified Rankin Scale ≥2 before onset
8. Use of tirofiban within 1 week before or after onset
9. Low platelets (<100×10^9 /L), or Prothrombin time >1.3 times of the upper normal limit, or INR >1.5, or other systemic hemorrhagic tendencies such as hematologic disorders
10. Elevation of ALT or AST more than 1.5 times the upper normal limit;
11. Glomerular filtration rate <60 ml/min/1.73m^2
12. Known malignant tumors
13. History of trauma or major surgical intervention within 6 weeks prior to onset
14. History of intracranial hemorrhage
15. Active or recent history(within 30 days prior to onset) of clinical bleeding (e.g., gastrointestinal bleeding)
16. Malignant hypertension (systolic blood pressure >200 mmHg, or diastolic blood pressure >120 mmHg)
17. Life expectancy ≤ 6 months
18. Contraindications of 3 T MRI examination
19. Pregnant or lactating women
20. Have participated in another clinical trial within 3 months prior to the date of informed consent, or are participating in another clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 516 (Actual)
Dates: Start 2023-11-09 (Actual); Primary Completion 2026-02-22 (Estimated); Study Completion 2026-03-20 (Estimated)

PRIMARY OUTCOMES:
Excellent functional outcome | 90 days
  Primary efficacy outcome: Excellent functional outcome is defined as modified Rankin Scale score: 0-1.
  Modified Rankin Scale, a commonly used scale for measuring the degree of dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. 0 - No symptoms.1 - No significant disability. Able to carry out all usual activities, despite some symptoms.2 - Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities.3 - Moderate disability. Requires some help, but able to walk unassisted.4 - Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted.5 - Severe disability. Requires constant nursing care and attention, bedridden, incontinent. 6 - Death.

SECONDARY OUTCOMES:
Excellent functional outcome | 7 days
  modified Rankin Scale score: 0-1
mRS | 7 and 90 days
  The modified Rankin Scale (mRS) is a commonly used 7-point ordinal scale ranging from 0 (no symptoms) to 6 (death), used to measure the degree of dependence in daily activities among patients with stroke or other neurological disabilities. The distribution of mRS scores at 7 and 90 days will be compared between the two study groups as an ordinal outcome, with higher scores indicating worse outcomes.
Early neurological deterioration | 7 days of randomization
  The presence of END is determined by an increase of ≥ 4 points in the NIHSS or an increase of ≥2 points in the NIHSS motor score. In addition, NIHSS motor score refers to bilateral upper and lower extremity mobility scores. The baseline NIHSS score for the calculation of END is the first clinician-evaluated and recorded NIHSS score after onset. The time frame for post-randomization END is within 7 days of randomization.
NIHSS score | 7 days and 90 days
  The NIHSS is a tool used by healthcare providers to objectively quantify the impairment caused by a stroke. The NIHSS is composed of 11 items, each of which scores a specific ability between a 0 and 4. For each item, a score of 0 typically indicates normal function in that specific ability, while a higher score is indicative of some level of impairment. The individual scores from each item are summed in order to calculate a patient's total NIHSS score. The maximum possible score is 42, with the minimum score being a 0.
Barthel index score | 90 days
  The Barthel Index (BI) is tool to measure the extent to which somebody can function independently and has mobility in activities of daily living (ADL), including 10 aspects: feeding, bathing, grooming, dressing, bowel control, bladder control, toileting, chair transfer, ambulation and stair climbing. Higher score indicates better performance in activities of daily living.
Ischemic stroke | 90 days
  Number of participants with new-onset ischemic stroke, confirmed by senior neurologists and the Clinical Event Committee.
Stroke | 90 days
  Number of participants with new-onset ischemic or hemorrhagic stroke, confirmed by senior neurologists and the Clinical Event Committee.
TIA | 90 days
  Number of participants with new-onset transient ischemic attack (TIA), confirmed by senior neurologists and the Clinical Event Committee.
Composite endpoint | 90 days
  Number of participants with new-onset stroke, myocardial Infarction, or all-cause death, confirmed by the Clinical Event Committee.
Proportion of Major bleeding | 7 days and 90 days
  Proportion of major bleeding defined by the PLATO criteria.
Serious adverse events | 90 days
  Serious adverse events
Adverse events | 90 days
  Adverse events
All-cause death | 90 days
  All-cause death
Changes in hemoglobin | 48 hours
  Blood test of the count of hemoglobin, g/L
Changes in the count of red blood cell | 48 hours
  Blood test of the count of red blood cell, 10^12/L
Changes in the count of white blood cell | 48 hours
  Blood test of the count of white blood cell, 10^9/L
Changes in the count of platelets | 48 hours
  Blood test of the count of platelets, 10^9/L
Changes in alanine transaminase | 48 hours
  Serum biochemical test for alanine transaminase
Changes in aspartate aminotransferase | 48 hours
  Serum biochemical test for aspartate aminotransferase
Changes in direct bilirubin | 48 hours
  Serum biochemical test for the concentration of direct bilirubin
Changes in indirect bilirubin | 48 hours
  Serum biochemical test for the concentration of indirect bilirubin
Changes in concentration of Na | 48 hours
  Serum biochemical test for the concentration of sodium, mmol/L
Changes in the concentration of K | 48 hours
  Serum biochemical test for the concentration of potassium, mmol/L
Changes in the concentration of creatinine | 48 hours
  Serum biochemical test for creatinine
Changes in the concentration of albumin | 48 hours
  Serum biochemical test for albumin
Changes in the urinary occult blood | 48 hours
  The test of urine blood (BLD). Negative or positive.
Changes in the fecal occult blood | 48 hours
  The test of occult blood (Occult blood, OB). Negative or positive

CONTACTS AND LOCATIONS:
Overall Officials: Jun Ni, MD, Principal Investigator — The office for BRANT study
Locations (25):
- China (25):
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Beijing Shunyi Hospital, Beijing, Beijing Municipality
  - Beijing Shijitan Hospital, Capital Medical University, Beijing, Beijing Municipality
  - The First Hospital of Tsinghua University, Beijing, Beijing Municipality
  - The second hospital of Baoding, Baoding, Hebei
  - Botou City Hospital, Botou, Hebei
  - Cangzhou Central Hospital, Cangzhou, Hebei
  - Chengde Central Hospital, Chengde, Hebei
  - Affiliated Hospital of Chifeng University, Chifeng, Hebei
  - Hengshui People's Hospital, Hengshui, Hebei
  - North China University of Science and Technology Affiliated Hospital, Tangshan, Hebei
  - The Second Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Yellow River SANMENXIA Hospital, Sanmenxia, Henan
  - The First People's Hospital of Shangqiu, Shangqiu, Henan
  - The First Affiliated Hospital of Xinxiang Medical Unversity, Xinxiang, Henan
  - Xuzhou Central Hospital, Xuzhou, Jiangsu
  - Meihekou Central Hospital, Meihekou, Jilin
  - Shengli Oilfield Central Hospital, Dongying, Shandong
  - Jinan Central Hospital, Jinan, Shandong
  - Deyang People's Hospital, Deyang, Sichuan
  - Mianyang Central Hospital, Mianyang, Sichuan
  - The First People's Hospital of Yibin, Yibin, Sichuan
  - The Second People's Hospital of Yibin, Yibin, Sichuan
  - The Second Hospital of Tianjin Medical University, Tianjing, Tianjing
  - Tibet Autonomous Region People's Hospital, Lhasa, Tibet

IPD SHARING:
Plan to Share IPD: Yes
The data that support the findings of this study are available from the corresponding author on reasonable request.

REFERENCES:
- [Background] Petrone L, Nannoni S, Del Bene A, Palumbo V, Inzitari D. Branch Atheromatous Disease: A Clinically Meaningful, Yet Unproven Concept. Cerebrovasc Dis. 2016;41(1-2):87-95. doi: 10.1159/000442577. Epub 2015 Dec 16. PMID 26671513
- [Background] Bang OY. Considerations When Subtyping Ischemic Stroke in Asian Patients. J Clin Neurol. 2016 Apr;12(2):129-36. doi: 10.3988/jcn.2016.12.2.129. Epub 2016 Jan 28. PMID 26833987
- [Background] Zhang C, Wang Y, Zhao X, Wang D, Liu L, Wang C, Pu Y, Zou X, Du W, Jing J, Pan Y, Wong KS, Wang Y; Chinese Intracranial Atherosclerosis Study Group. Distal single subcortical infarction had a better clinical outcome compared with proximal single subcortical infarction. Stroke. 2014 Sep;45(9):2613-9. doi: 10.1161/STROKEAHA.114.005634. Epub 2014 Jul 22. PMID 25052317
- [Background] Jeong HG, Kim BJ, Yang MH, Han MK, Bae HJ. Neuroimaging markers for early neurologic deterioration in single small subcortical infarction. Stroke. 2015 Mar;46(3):687-91. doi: 10.1161/STROKEAHA.114.007466. Epub 2015 Feb 12. PMID 25677600
- [Background] Seners P, Ben Hassen W, Lapergue B, Arquizan C, Heldner MR, Henon H, Perrin C, Strambo D, Cottier JP, Sablot D, Girard Buttaz I, Tamazyan R, Preterre C, Agius P, Laksiri N, Mechtouff L, Bejot Y, Duong DL, Mounier-Vehier F, Mione G, Rosso C, Lucas L, Papassin J, Aignatoaie A, Triquenot A, Carrera E, Niclot P, Obadia A, Lyoubi A, Garnier P, Crainic N, Wolff V, Tracol C, Philippeau F, Lamy C, Soize S, Baron JC, Turc G; MINOR-STROKE Collaborators. Prediction of Early Neurological Deterioration in Individuals With Minor Stroke and Large Vessel Occlusion Intended for Intravenous Thrombolysis Alone. JAMA Neurol. 2021 Mar 1;78(3):321-328. doi: 10.1001/jamaneurol.2020.4557. PMID 33427887
- [Background] Duan Z, Fu C, Chen B, Xu G, Tao L, Tang T, Hou H, Fu X, Yang M, Liu Z, Zhang X. Lesion patterns of single small subcortical infarct and its association with early neurological deterioration. Neurol Sci. 2015 Oct;36(10):1851-7. doi: 10.1007/s10072-015-2267-1. Epub 2015 Jun 2. PMID 26032577
- [Background] Helleberg BH, Ellekjaer H, Indredavik B. Outcomes after Early Neurological Deterioration and Transitory Deterioration in Acute Ischemic Stroke Patients. Cerebrovasc Dis. 2016;42(5-6):378-386. doi: 10.1159/000447130. Epub 2016 Jun 29. PMID 27351585
- [Background] Heitsch L, Ibanez L, Carrera C, Binkley MM, Strbian D, Tatlisumak T, Bustamante A, Ribo M, Molina C, Davalos A, Lopez-Cancio E, Munoz-Narbona L, Soriano-Tarraga C, Giralt-Steinhauer E, Obach V, Slowik A, Pera J, Lapicka-Bodzioch K, Derbisz J, Sobrino T, Castillo J, Campos F, Rodriguez-Castro E, Arias-Rivas S, Segura T, Serrano-Heras G, Vives-Bauza C, Diaz-Navarro R, Tur S, Jimenez C, Marti-Fabregas J, Delgado-Mederos R, Arenillas J, Krupinski J, Cullell N, Torres-Aguila NP, Muino E, Carcel-Marquez J, Moniche F, Cabezas JA, Ford AL, Dhar R, Roquer J, Khatri P, Jimenez-Conde J, Fernandez-Cadenas I, Montaner J, Rosand J, Cruchaga C, Lee JM; International Stroke Genetics Consortium. Early Neurological Change After Ischemic Stroke Is Associated With 90-Day Outcome. Stroke. 2021 Jan;52(1):132-141. doi: 10.1161/STROKEAHA.119.028687. Epub 2020 Dec 15. PMID 33317415
- [Background] Park MG, Oh EH, Kim BK, Park KP. Intravenous tissue plasminogen activator in acute branch atheromatous disease: Does it prevent early neurological deterioration? J Clin Neurosci. 2016 Nov;33:194-197. doi: 10.1016/j.jocn.2016.04.011. Epub 2016 Jul 21. PMID 27452127
- [Background] Seners P, Turc G, Oppenheim C, Baron JC. Incidence, causes and predictors of neurological deterioration occurring within 24 h following acute ischaemic stroke: a systematic review with pathophysiological implications. J Neurol Neurosurg Psychiatry. 2015 Jan;86(1):87-94. doi: 10.1136/jnnp-2014-308327. Epub 2014 Jun 26. PMID 24970907
- [Background] Ospel JM, Menon BK, Demchuk AM, Almekhlafi MA, Kashani N, Mayank A, Fainardi E, Rubiera M, Khaw A, Shankar JJ, Dowlatshahi D, Puig J, Sohn SI, Ahn SH, Poppe A, Calleja A, Hill MD, Goyal M. Clinical Course of Acute Ischemic Stroke Due to Medium Vessel Occlusion With and Without Intravenous Alteplase Treatment. Stroke. 2020 Nov;51(11):3232-3240. doi: 10.1161/STROKEAHA.120.030227. Epub 2020 Oct 19. PMID 33070714
- [Background] Wu X, Liu Y, Nie C, Kang Z, Wang Q, Sun D, Li H, Liu Y, Mei B. Efficacy and Safety of Intravenous Thrombolysis on Acute Branch Atheromatous Disease: A Retrospective Case-Control Study. Front Neurol. 2020 Jul 7;11:581. doi: 10.3389/fneur.2020.00581. eCollection 2020. PMID 32733357
- [Background] Yi X, Zhou Q, Wang C, Lin J, Chai Z. Aspirin plus clopidogrel may reduce the risk of early neurologic deterioration in ischemic stroke patients carrying CYP2C19*2 reduced-function alleles. J Neurol. 2018 Oct;265(10):2396-2403. doi: 10.1007/s00415-018-8998-1. Epub 2018 Aug 20. PMID 30128710
- [Background] Yi X, Zhou Q, Zhang Y, Zhou J, Lin J. Variants in clopidogrel-relevant genes and early neurological deterioration in ischemic stroke patients receiving clopidogrel. BMC Neurol. 2020 Apr 28;20(1):159. doi: 10.1186/s12883-020-01703-6. PMID 32345264
- [Background] Wang Q, Chen C, Chen XY, Han JH, Soo Y, Leung TW, Mok V, Wong KS. Low-molecular-weight heparin and early neurologic deterioration in acute stroke caused by large artery occlusive disease. Arch Neurol. 2012 Nov;69(11):1454-60. doi: 10.1001/archneurol.2012.1633. PMID 22893265
- [Background] Yang J, Wu Y, Gao X, Bivard A, Levi CR, Parsons MW, Lin L; INSPIRE Study Groupdagger. Intraarterial Versus Intravenous Tirofiban as an Adjunct to Endovascular Thrombectomy for Acute Ischemic Stroke. Stroke. 2020 Oct;51(10):2925-2933. doi: 10.1161/STROKEAHA.120.029994. Epub 2020 Sep 16. PMID 32933416
- [Background] Wu C, Sun C, Wang L, Lian Y, Xie N, Huang S, Zhao W, Ren M, Wu D, Ding J, Song H, Wang Y, Ma Q, Ji X. Low-Dose Tirofiban Treatment Improves Neurological Deterioration Outcome After Intravenous Thrombolysis. Stroke. 2019 Dec;50(12):3481-3487. doi: 10.1161/STROKEAHA.119.026240. Epub 2019 Oct 1. PMID 31570084
- [Background] Liu B, Zhang H, Wang R, Qu H, Sun Y, Zhang W, Zhang S. Early administration of tirofiban after urokinase-mediated intravenous thrombolysis reduces early neurological deterioration in patients with branch atheromatous disease. J Int Med Res. 2020 May;48(5):300060520926298. doi: 10.1177/0300060520926298. PMID 32459110
- [Background] Pan X, Zheng D, Zheng Y, Chan PWL, Lin Y, Zou J, Zhou J, Yang J. Safety and efficacy of tirofiban combined with endovascular treatment in acute ischaemic stroke. Eur J Neurol. 2019 Aug;26(8):1105-1110. doi: 10.1111/ene.13946. Epub 2019 Mar 19. PMID 30793464
- [Background] Chung JW, Kim BJ, Sohn CH, Yoon BW, Lee SH. Branch atheromatous plaque: a major cause of lacunar infarction (high-resolution MRI study). Cerebrovasc Dis Extra. 2012 Jan;2(1):36-44. doi: 10.1159/000341399. Epub 2012 Jul 27. PMID 23060895
- [Background] Liang J, Liu Y, Xu X, Shi C, Luo L. Cerebral Perforating Artery Disease : Characteristics on High-Resolution Magnetic Resonance Imaging. Clin Neuroradiol. 2019 Sep;29(3):533-541. doi: 10.1007/s00062-018-0682-4. Epub 2018 Mar 23. PMID 29572675
- [Background] Liao S, Deng Z, Wang Y, Jiang T, Kang Z, Tan S, Shan Y, Zou Y, Lu Z. Different Mechanisms of Two Subtypes of Perforating Artery Infarct in the Middle Cerebral Artery Territory: A High-Resolution Magnetic Resonance Imaging Study. Front Neurol. 2018 Sep 20;9:657. doi: 10.3389/fneur.2018.00657. eCollection 2018. PMID 30294295
- [Background] Zhao DL, Deng G, Xie B, Gao B, Peng CY, Nie F, Yang M, Ju S, Teng GJ. Wall characteristics and mechanisms of ischaemic stroke in patients with atherosclerotic middle cerebral artery stenosis: a high-resolution MRI study. Neurol Res. 2016 Jul;38(7):606-13. doi: 10.1179/1743132815Y.0000000088. Epub 2016 May 9. PMID 26315990
- [Background] Wallentin L, Becker RC, Budaj A, Cannon CP, Emanuelsson H, Held C, Horrow J, Husted S, James S, Katus H, Mahaffey KW, Scirica BM, Skene A, Steg PG, Storey RF, Harrington RA; PLATO Investigators; Freij A, Thorsen M. Ticagrelor versus clopidogrel in patients with acute coronary syndromes. N Engl J Med. 2009 Sep 10;361(11):1045-57. doi: 10.1056/NEJMoa0904327. Epub 2009 Aug 30. PMID 19717846
- [Background] Hansson L, Hedner T, Dahlof B. Prospective randomized open blinded end-point (PROBE) study. A novel design for intervention trials. Prospective Randomized Open Blinded End-Point. Blood Press. 1992 Aug;1(2):113-9. doi: 10.3109/08037059209077502. PMID 1366259
- [Derived] Li S, Zhang D, Sha Y, Zhu Y, Zhou L, Peng B, Ni J. Efficacy and safety of tirofiban in patients with acute branch atheromatous disease-related stroke (BRANT): a protocol for a randomised controlled trial. BMJ Open. 2024 Jun 10;14(6):e082141. doi: 10.1136/bmjopen-2023-082141. PMID 38858147
- See also: Zhou LX, Ni J.Advances in Branch Atheromatous Disease. Chinese Stroke Journal 2020;15:1342- 1351 — http://www.wanfangdata.com.cn/details/detail.do?_type=perio&id=zgzzzz202012015
- See also: Chinese Stroke Association. Expert consensus on the clinical application of tirofiban in atherosclerotic cerebrovascular disease. Chinese Stroke Journal 2019;14:1034- 1044 — http://www.wanfangdata.com.cn/details/detail.do?_type=perio&id=zgzzzz201910013
- See also: Chinese Society of Neurology, Cerebrovascular disease group of Chinese Society of Neurology. Chinese guidelines for diagnosis and treatment of acute ischemic stroke 2018. Chin J Neurol. 2018;51 9:666-82 — http://www.wanfangdata.com.cn/details/detail.do?_type=perio&id=zhsjk201809005